CLINICAL TRIAL: NCT02705638
Title: Treatment of IgG4-Related Disease With Revlimid and Rituximab: The TIGR2 Trial
Brief Title: Treatment of IgG4-Related Disease With Revlimid and Rituximab
Acronym: TIGR2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Thomas E. Witzig, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-003700
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Immunoglobulin G Subclass 4 Related Disease; IgG4-related Disease; Autoimmune Pancreatitis; IgG4-related Sclerosing Cholangitis; Retroperitoneal Fibrosis
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; Autoimmune Pancreatitis; Retroperitoneal Fibrosis | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab and Lenalidomide (Experimental): All subjects will receive Rituxan 1,000 mg intravenously on days 1 and 15, as well as Revlimid 20 mg orally per day on days 1-21, 29-49, and 57-77.
  Interventions: Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rituximab — All subjects will receive Rituxan 1,000 mg intravenously on days 1 and 15.
  Other Names: Rituxan
Drug: Lenalidomide — All subjects will receive Revlimid 20 mg orally per day on days 1-21, 29-49, and 57-77.
  Other Names: Revlimid

SUMMARY:
Among persons with Immunoglobulin G subclass 4 Related Disease (IgG4)-related disease who have persistent or recurrent disease despite standard therapies, does combination therapy with rituximab and revlimid cause a sustained disease remission?

DETAILED DESCRIPTION:
Immunoglobulin G subclass 4 Related Disease (IgG4-RD) is a recently recognized systemic fibroinflammatory condition. Various manifestations of IgG4-RD were previously recognized in individual organ systems, but these entities (including autoimmune pancreatitis, orbital pseudotumor, Reidel's thyroiditis, retroperitoneal fibrosis, idiopathic sialadenitis and dacryoadenitis, etc) are now recognized as manifestations of a common disease process that can affect any organ system. IgG4-RD is characterized by distinctive histologic findings of tissue infiltration by IgG4-positive plasma cells together with storiform fibrosis and obliterative phlebitis. Both clinical and pathologic consensus diagnostic criteria have been defined. Serum IgG4 concentration is a biomarker for IgG4-RD and is elevated in 70% to 90% of patients with active disease.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of active IgG4-RD based on standard pathologic or clinical criteria (see below) and requiring medical treatment
2. Patient is:

   1. in relapse after prior steroid and/or rituximab (RTX) treatment or while tapering steroid treatment, OR
   2. has disease that is refractory to steroids, OR
   3. has contraindications to steroid therapy (including diabetes, mood disorder, obesity)
3. Absolute neutrophil count >1500 and platelet count >/= 100,000
4. Calculated creatinine clearance (or estimated GFR) greater than or equal to 60ml/min
5. In patients without hepatobiliary involvement by IgG4-RD, total bilirubin less than or equal to 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) less than or equal to 3 x ULN
6. Not pregnant or nursing
7. All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS™) program, and be willing and able to comply with the requirements of the REMS™ program
8. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS™ program
9. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin)
10. Agrees to use acceptable methods of birth control during and for 12 months after completion of study drug therapy (applies to all men, and women of child bearing potential)
11. Females must follow pregnancy testing requirements as outlined in the Revlimid REMS™ program

Exclusion criteria:

1. Predominant changes of fibrosis (as opposed to active cellular inflammation) within the organs affected by IgG4-RD, such that the likelihood of a disease response to treatment is low
2. Presence of active infection that would interfere with therapy on this study, including positive serum hepatitis B surface antigen, HIV or active hepatitis C virus (HCV) infection, untreated syphilis or tuberculosis, clinical history of multiple herpes virus reactivations
3. Known immunodeficiency state
4. New York Heart Association Classification III or IV heart disease
5. Active malignancy requiring therapy
6. Receipt of a live vaccine within 4 weeks prior to initiating study drug therapy.
7. Allergies: History of severe allergic reactions to human or chimeric monoclonal antibodies, murine protein, or lenalidomide
8. Substance abuse: Drug or alcohol abuse that could interfere with participation in the trial according to the protocol
9. Known anti-human anti-chimeric antibody formation
10. Treatment with infliximab, adalimumab, or etanercept within the past 12 months.
11. Currently taking azathioprine, 6-mercaptopurine, methotrexate, mycophenolate mofetil, or other conventional immunomodulators. Patients receiving these drugs must discontinue them prior to enrollment
12. Other investigational medication within the previous one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects in remission for Immunoglobulin G subclass 4 Related Disease at 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Topazian, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No